CLINICAL TRIAL: NCT03528551
Title: Safety and Efficacy of Turoctocog Alfa Pegol (N8-GP) in Prophylaxis and Treatment of Bleeds in Previously N8-GP Treated Patients With Severe Haemophilia A
Brief Title: A Research Study Looking at How a Factor VIII Medicine Called Turoctocog Alfa Pegol (N8-GP) Works in People With Haemophilia A
Acronym: pathfinder8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7088-4410; U1111-1202-2780 (Other: World Health Organization (WHO)); 2017-003788-36 (Registry Identifier: European Medicines Agency (EudraCT)); JapicCTI-183952 (Registry Identifier: JAPIC)
Record Dates: First submitted 2018-04-18; First posted 2018-05-18 (Actual); Results first posted 2021-11-26 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- N8-GP, once weekly (Experimental): All participants will receive turoctocog alfa pegol (N8-GP) once weekly.
  Interventions: Drug: Turoctocog alfa pegol
- N8-GP, twice weekly (Experimental): All participants will receive N8-GP twice weekly.
  Interventions: Drug: Turoctocog alfa pegol
- N8-GP, three times weekly (Experimental): All participants will receive N8-GP three times weekly.
  Interventions: Drug: Turoctocog alfa pegol

INTERVENTIONS:
Drug: Turoctocog alfa pegol — Turoctocog alfa pegol 75 IU/kg body weight will be administered once weekly as intravenous injections for a duration of 2 years.
  Arms: N8-GP, once weekly
Drug: Turoctocog alfa pegol — Turoctocog alfa pegol 60 IU/kg body weight (for patients younger than 12 years) and 50 IU/kg body weight (for patients, 12 years or older) will be administered twice weekly as intravenous injections for a duration of 2 years.
  Arms: N8-GP, twice weekly
Drug: Turoctocog alfa pegol — Turoctocog alfa pegol 50 IU/kg body weight will be administered three times weekly as intravenous injections for a duration of 2 years.
  Arms: N8-GP, three times weekly

SUMMARY:
This study will look at how a known study medicine N8-GP works in previously N8-GP treated people with haemophilia A. The aim is to look at how N8-GP works during regular use. Participants will get N8-GP. N8-GP has been tested in more than 200 people with haemophilia A for several years. Participants will get an injection of N8-GP into a blood vessel, one, two or three times weekly. Participants will get more doses if they bleed or if they will need a surgery. The study will last for about 2 years. Participants will have at least 9 visits with the study doctor. If participants agree to be in this study, they will get their first injection (in this study) at the first visit. Participants will also get an injection at visit 3, 5 and 7. Participants will be trained to give all other injections themselves. Participants must not use any clotting factors other than N8-GP or any anticoagulants (blood thinners) during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male patients of all ages with the diagnosis of severe congenital haemophilia A (coagulation Factor VIII [FVIII] activity less than 1%) based on medical records
* On-going participation in NN7088-3859 (pathfinder2), or NN7088-3885 (pathfinder5) at the time of transfer

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product including allergy to hamster protein or related products
* Any disorder, except for conditions associated with haemophilia, which in the investigator's opinion might jeopardise patient's safety or compliance with the protocol - Current participation in any clinical trial (except NN7088-3859 (pathfinder2) or NN7088-3885 (pathfinder5)) of an approved or non-approved investigational medicinal product

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure 2834, Study Director — Novo Nordisk A/S
Locations (64):
- United States (18):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, East Lansing, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, New Hyde Park, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Norfolk, Virginia
- Australia (2):
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, Parkville, Victoria
- Novo Nordisk Investigational Site, Campinas, São Paulo, Brazil
- Novo Nordisk Investigational Site, Toronto, Ontario, Canada
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Novo Nordisk Investigational Site, Århus N, Denmark
- France (3):
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Nantes
- Germany (3):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Frankfurt/M.
  - Novo Nordisk Investigational Site, Homburg
- Novo Nordisk Investigational Site, Athens, Greece
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Italy (2):
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Vicenza
- Japan (3):
  - Novo Nordisk Investigational Site, Kitakyusyu-shi, Fukuoka
  - Novo Nordisk Investigational Site, Nara
  - Novo Nordisk Investigational Site, Tokyo
- Novo Nordisk Investigational Site, Vilnius, Lithuania
- Novo Nordisk Investigational Site, Selangor Darul Ehsan, Malaysia
- Netherlands (2):
  - Novo Nordisk Investigational Site, Groningen
  - Novo Nordisk Investigational Site, Rotterdam
- Novo Nordisk Investigational Site, Oslo, Norway
- Novo Nordisk Investigational Site, Porto, Portugal
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Novo Nordisk Investigational Site, Daejeon, South Korea
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
- Switzerland (3):
  - Novo Nordisk Investigational Site, Bellinzona
  - Novo Nordisk Investigational Site, Lausanne
  - Novo Nordisk Investigational Site, Zurich
- Novo Nordisk Investigational Site, Taipei, Taiwan
- Turkey (Türkiye) (5):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, İzmit
  - Novo Nordisk Investigational Site, Samsun
- Novo Nordisk Investigational Site, Lviv, Ukraine
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Basingstoke
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 66 sites in 25 countries: Australia(2), Brazil(1), Canada(1), Croatia(1), Denmark(1), France(2), Germany(2), Greece(1), Hungary(2), Israel(1), Italy(2), Japan(3), Korea(1), Lithuania(1), Malaysia(1), Netherlands(2), Norway(1), Portugal(1), Spain(2), Switzerland(4), Taiwan(1), Turkey(5), Ukraine(1), United Kingdom (8), United States (USA) (19).
Pre-assignment Details: Out of 160 participants enrolled in this study, 102 came from trial NN7088-3859 and 58 came from trial NN7088-3885. The participants received turoctocog alfa pegol (N8-GP) injections either as once-weekly, twice weekly or three times weekly during the 104 weeks treatment period. Despite 160 participants started the trial, the total number of participants considered are 167 as 2 participants switched to twice weekly and 5 participants switched to three times weekly regimen.
Groups:
- N8-GP, Once Weekly: Participants received once weekly (dosing every 7 day) prophylaxis doses of N8-GP, 75 IU/kg (International Units per kilogram) intravenous injections for 104 weeks. Participants treated with N8-GP once weekly or were on the on demand regimen in the previous trial NN7088-3859 (pathfinder2) were included in this arm. At the investigator's discretion an intensification of the dosing regimen to twice weekly was allowed if the participant experienced more than 2 bleeds within an 8 week period or experienced a severe bleed requiring hospitalization.
- N8-GP, Twice Weekly: Participants received twice weekly (dosing every 3 and 4 days) prophylaxis doses of N8-GP intravenous injections for 104 weeks: N8-GP, 50 IU/kg for participants aged ≥ 12 years and N8-GP, 60 IU/kg for participants aged < 12 years. Participants treated with N8-GP in the previous trials NN7088-3859 (pathfinder2) and NN7088-3885 (pathfinder5) were included in this arm. At the investigator's discretion, an intensification of the dosing regimen to thrice weekly was allowed if the participant experienced spontaneous bleeding episodes. Participants in this arm were permitted to switch to three times weekly at any time if clinically justified. Otherwise any treatment regimen was preferably be kept for a minimum of 6 months.
- N8-GP, Three Times Weekly: Participants received three times weekly (dosing every 2, 2 and 3 days) prophylaxis doses of N8-GP, 50 IU/kg as intravenous injections for a duration of 104 weeks. Participants treated with N8-GP in the previous trials NN7088-3859 (pathfinder2) and NN7088-3885 (pathfinder5) were included in this arm. Participants in this arm were permitted to switch to twice weekly at any time if clinically justified. Otherwise any treatment regimen was preferably be kept for a minimum of 6 months.
Period: Overall Study
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Started | 25 | 133 | 2
Completed | 23 | 114 | 2
Not Completed | 2 | 19 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Transferred to other arm/group | 2 | 3 | 0
Not completed — Withdrawal by parent/guardian | 0 | 5 | 0
Not completed — Protocol Violation | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 7 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants exposed to at least one dose of trial product in the current trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly | Total
Number analyzed (Participants) | 25 | 133 | 2 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.1 (12.7) | 27.3 (16.8) | 25.3 (17.8) | 28.4 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 25 | 133 | 2 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 8 | 0 | 8
  Not Hispanic or Latino | 25 | 124 | 2 | 151
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 17 | 1 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 0 | 5
  White | 21 | 108 | 1 | 130
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Reported
Description: An adverse event (AE) was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All AEs mentioned here are treatment emergent adverse events (TEAEs). The TEAE is defined as an event reported from date of first trial product administration until end of the treatment visit (week 104) or follow-up visit if relevant (1 month after end of the treatment).
Time Frame: Week 0 to week 108
Population: Safety analysis set (SAS) included all enrolled participants who were exposed to the trial product.
Measure: Number; unit: Events
Groups:
- N8-GP, Twice Weekly: Participants received twice weekly (dosing every 3 and 4 days) prophylaxis doses of N8-GP intravenous injections for 104 weeks: N8-GP, 50 IU/kg for participants aged ≥ 12 years and N8-GP, 60 IU/kg for participants aged < 12 years. Participants treated with N8-GP in the previous trials NN7088-3859 (pathfinder2) and NN7088-3885 (pathfinder5) were included in this arm. At the investigator's discretion, an intensification of the dosing regimen to thrice weekly was allowed if the participant experienced spontaneous bleeding episodes. Participants in this arm were permitted to switch to three times weekly at any time if clinically justified. Otherwise any treatment regimen was preferably be kept for a minimum of 6 months. During the trial, 2 participants switched from once weekly to twice weekly regimen for treatment intensification. Thus, though 133 participants have started the trial with twice weekly regimen, the data is presented for 135 participants in this arm (i.e. 133+2 = 135).
- N8-GP, Three Times Weekly: Participants received three times weekly (dosing every 2, 2 and 3 days) prophylaxis doses of N8-GP, 50 IU/kg as intravenous injections for a duration of 104 weeks. Participants treated with N8-GP in the previous trials NN7088-3859 (pathfinder2) and NN7088-3885 (pathfinder5) were included in this arm. Participants in this arm were permitted to switch to twice weekly at any time if clinically justified. Otherwise any treatment regimen was preferably be kept for a minimum of 6 months. During the trial, 5 participants switched from twice weekly to three times weekly regimen for treatment intensification. Thus, though 2 participants have started the trial with three times regimen, the data is presented for 7 participants in this arm (i.e. 2+5 = 7).
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 25 | 135 | 7
Events | 58 | 444 | 8

2. Secondary Outcome: Number of Participants With Inhibitory Antibodies Against Coagulation Factor VIII (FVIII) ≥0.6 Bethesda Units (BU)
Description: The Incidence of inhibitors against coagulation factor eight (FVIII) is defined as titre greater than or equal to (≥) 0.6 Bethesda unit. The inhibitor antibodies were measured using a heat modified Nijmegen FVIII Bethesda assay. The number of participants who developed inhibitors against FVIII are reported.
Time Frame: Week 0 to week 104
Population: FAS included all participants exposed to at least one dose of trial product in the current trial.
Measure: Number; unit: Participants
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 25 | 135 | 7
Participants | 0 | 0 | 0

3. Secondary Outcome: Number of Bleeding Episodes on Prophylaxis
Description: Number of bleeding episodes per participant in the prophylaxis regimen was evaluated during 104 weeks.
Time Frame: Week 0 to week 104
Population: FAS included all participants exposed to at least one dose of trial product in the current trial.
Measure: Number; unit: Episodes
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 25 | 135 | 7
Episodes | 123 | 190 | 14

4. Secondary Outcome: Number of Spontaneous Bleeding Episodes on Prophylaxis
Description: Spontaneous bleeding referred as bleeding episodes that occurred without apparent cause. The number of spontaneous bleeding episodes were evaluated during 104 weeks.
Time Frame: Week 0 to week 104
Population: FAS included all participants exposed to at least one dose of trial product in the current trial.
Measure: Number; unit: Episodes
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 25 | 135 | 7
Episodes | 98 | 73 | 8

5. Secondary Outcome: Haemostatic Effect of N8-GP When Used for Treatment of Bleeding Episodes Assessed as: Excellent, Good, Moderate, or None
Description: The haemostatic effect after treatment of a bleed with N8-GP was assessed using a 4-point scale: 'excellent', 'good', 'moderate' or 'none'. The evaluation was done as follows: 1. Excellent: Abrupt pain relief and/or unequivocal improvement in objective signs of bleeding within approximately 8 hours after a single injection. 2. Good: Definite pain relief and/or improvement in signs of bleeding within approximately 8 hours after an injection, but possibly requiring more than one injection for complete resolution. 3. Moderate: Probable or slight beneficial effect within approximately 8 hours after the first injection; usually requiring more than one injection 4. None: No improvement or worsening of symptoms.
Time Frame: Week 0 to week 104
Population: FAS included all participants exposed to at least one dose of trial product in the current trial.
Measure: Number; unit: Episodes
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 25 | 135 | 7
Episodes
  Excellent | 114 | 94 | 8
  Good | 8 | 80 | 6
  Moderate | 0 | 4 | 0
  None | 0 | 0 | 0
  Missing | 0 | 8 | 0

6. Secondary Outcome: Mean Number of N8-GP Injections Required Per Bleeding Episode
Description: The mean number of N8-GP injections required per bleeding episode from start to stop of a bleed for participants was presented from week 0 to week 104.
Time Frame: Week 0 to week 104
Population: FAS included all participants exposed to at least one dose of trial product in the current trial.
Measure: Mean (Standard Deviation); unit: Injections per bleed
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 25 | 135 | 7
Injections per bleed | 1.2 (0.6) | 1.5 (1.3) | 1.1 (0.4)

7. Secondary Outcome: Pre-dose FVIII Activity Levels on N8-GP Prophylaxis
Description: The pre-dose FVIII activity levels were assessed in International units per millilitre (IU/mL) units from week 0 to week 104 to get an estimate of the pre-dose level for N8-GP at steady-state using mixed model.
Time Frame: Week 0 to week 104
Population: FAS included all participants exposed to at least one dose of trial product in the current trial.
Measure: Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 25 | 135 | 7
IU/mL | 0.016 [0.011 to 0.023] | 0.042 [0.035 to 0.049] | 0.049 [0.018 to 0.133]

8. Secondary Outcome: Change in Joint Health Status From Start to End of Trial (Based on Haemophilia Joint Health Score)
Description: Haemophilia Joint Health Score is a validated outcome tool developed for the assessment of joint health in patients with hemophilia. It comprises an evaluation of the elbow, knee and ankle joints with regards to swelling, muscular atrophy, crepitation and range of motion, joint pain, strength, motion and axial alignment. The score range is from 0 to 24 points (a score of 0 indicates no joint damage. Higher the score higher the joint damage). Change from week 0 to end of trial (week 104) in the domain scores was presented.
Time Frame: Week 0, Week 104
Population: FAS included all participants exposed to at least one dose of trial product in the current trial. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 21 | 112 | 2
Score on a scale | 0.238 (7.75) | -0.116 (7.40) | -10.0 (14.1)

9. Secondary Outcome: Haemostatic Response During Major Surgical Interventions Assessed as: Excellent, Good, Moderate, or None
Description: The Haemostatic response to N8-GP during major surgical interventions was assessed using a 4-point scale: 'excellent', 'good', 'moderate' or 'none'. The evaluation was done as follows: 1. Excellent: Better than expected/predicted in this type of procedure. 2. Good: As expected in this type of procedure 3. Moderate: Less than optimal for the type of procedure but haemostatic response maintained without change of treatment regimen 4. None: Bleeding due to inadequate therapeutic response with adequate dosing, change of regimen required. This endpoint was measured from week 0 to week 104.
Time Frame: Week 0 to week 104
Population: FAS included all participants exposed to at least one dose of trial product in the current trial.
Measure: Number; unit: Surgeries
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 25 | 135 | 7
Surgeries
  Excellent | 3 | 8 | 0
  Good | 1 | 4 | 0
  Moderate | 0 | 0 | 0
  None | 0 | 0 | 0
  Missing | 0 | 1 | 0

10. Secondary Outcome: Consumption of N8-GP Per Bleed
Description: The average dose of N8-GP consumed for treatment of bleed was assessed in International units per kilogram per bleed(IU/kg/bleed). This endpoint was evaluated from week 0 to week 104.
Time Frame: Week 0 to week 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: IU/kg/bleed
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 10 | 61 | 3
IU/kg/bleed | 91.3 (85.0) | 81.9 (55.9) | 61.1 (12.0)

11. Secondary Outcome: Consumption of N8-GP During Prophylaxis Treatment
Description: The average dose of N8-GP consumed for prevention of bleed was assessed. This endpoint was evaluated from week 0 to week 104.
Time Frame: Week 0 to week 104
Population: FAS included all participants exposed to at least one dose of trial product in the current trial.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 25 | 135 | 7
IU/kg | 3878 (296.4) | 5320 (565.0) | 7646 (877.2)

12. Secondary Outcome: Change From Start Till End of Trial in Treatment Satisfaction (Based on Hemo-SAT Score)
Description: The treatment satisfaction of a bleed with N8-GP was assessed using HEMO-SAT assessment tool which contains a questionnaire with 6 domains (Ease and convenience, efficacy, burden, specialist/nurses, centre/hospital, general satisfaction), with a scale of 0-100. The lower scores reflecting greater treatment satisfaction. In other words, decrease in the score would mean improvement. The summary of change presented was based on individual changes since week 0. Data is presented for total score.
Time Frame: Week 0, Week 104
Population: FAS included all participants exposed to at least one dose of trial product in the current trial. 'Overall Number of Participants Analyzed' = participants with available data. Number analysed = Number of participants who contributed to the analysis. In the N8-GP, once weekly arm; none of the subjects were aged <=16 years. Hence the number analyzed is mentioned as zero.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly
Number analyzed (Participants) | 23 | 118 | 7
Score on a scale
  Total Score (participants aged >= 17 years): number analyzed (Participants) | 23 | 73 | 3
  Total Score (participants aged >= 17 years) | -4.65 (8.16) | -2.11 (7.48) | -12.3 (23.78)
  Total Score (participants aged <=16 years): number analyzed (Participants) | 0 | 45 | 4
  Total Score (participants aged <=16 years) |  | -1.78 (8.54) | 1.43 (7.31)

ADVERSE EVENTS:
Time Frame: Week 0 to week 108
Description: All adverse events are treatment emergent (TEAEs). The TEAEs were defined as the events reported from date of first trial product administration until end of the treatment visit (week 104) or follow-up visit if relevant (1 month after end of the treatment). SAS included all enrolled participants as they were previously been exposed to trial product.
Groups:
- N8-GP, Twice Weekly: Participants received twice weekly (dosing every 3 and 4 days) prophylaxis doses of N8-GP intravenous injections for 104 weeks: N8-GP, 50 IU/kg for participants aged ≥ 12 years and N8-GP, 60 IU/kg for participants aged < 12 years. Participants treated with N8-GP in the previous trials NN7088-3859 (pathfinder2) and NN7088-3885 (pathfinder5) were included in this arm. At the investigator's discretion, an intensification of the dosing regimen to thrice weekly was allowed if the participant experienced spontaneous bleeding episodes. Participants in this arm were permitted to switch to three times weekly at any time if clinically justified. Otherwise any treatment regimen was preferably be kept for a minimum of 6 months. During the trial, 2 participants switched from once weekly to twice weekly regimen for treatment intensification. Thus, though 133 participants have started the trial with twice weekly regimen, AE data is presented for 135 participants in this arm (i.e. 133+2 = 135).
- N8-GP, Three Times Weekly: Participants received three times weekly (dosing every 2, 2 and 3 days) prophylaxis doses of N8-GP, 50 IU/kg as intravenous injections for a duration of 104 weeks. Participants treated with N8-GP in the previous trials NN7088-3859 (pathfinder2) and NN7088-3885 (pathfinder5) were included in this arm. Participants in this arm were permitted to switch to twice weekly at any time if clinically justified. Otherwise any treatment regimen was preferably be kept for a minimum of 6 months. During the trial, 5 participants switched from twice weekly to three times weekly regimen for treatment intensification. Thus, though 2 participants have started the trial with three times regimen, AE data is presented for 7 participants in this arm (i.e. 2+5 = 7).
- Total: Total number of participants
Arm/Group | N8-GP, Once Weekly | N8-GP, Twice Weekly | N8-GP, Three Times Weekly | Total
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/135 | 0/7 | 1/160
Serious Adverse Events (participants affected / at risk) | 4/25 | 15/135 | 0/7 | 19/160
Other Adverse Events (participants affected / at risk) | 9/25 | 46/135 | 4/7 | 56/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N8-GP, Once Weekly (N=25) | N8-GP, Twice Weekly (N=135) | N8-GP, Three Times Weekly (N=7) | Total (N=160)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mole excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N8-GP, Once Weekly (N=25) | N8-GP, Twice Weekly (N=135) | N8-GP, Three Times Weekly (N=7) | Total (N=160)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 11 (12) | 1 (1) | 14 (15)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 0 (0) | 10 (11) | 0 (0) | 10 (11)
Influenza (Infections and infestations) | 0 (0) | 9 (9) | 0 (0) | 9 (9)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 21 (23) | 0 (0) | 24 (26)
Upper respiratory tract infection (Infections and infestations) | 4 (13) | 11 (18) | 1 (2) | 16 (33)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT03528551/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT03528551/SAP_001.pdf